CLINICAL TRIAL: NCT07067931
Title: The Effect of Stroboscopic Vision-Assisted Exercise Training on Ankle Muscle Architecture in Chronic Ankle Instability Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Medipol
Record Dates: First submitted 2025-07-06; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Chronic Ankle Instability; Muscle Architecture
Keywords: chronic ankle instabilty; stroboscopic vision; muscle architecture; piliometric
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The non-stroboscopic group (Experimental): The non-stroboscopic group will perform the exercises without glasses. The exercise training groups will follow an 8-week program, two sessions per week, involving combined balance and plyometric exercises. Plyometric training emphasizes the stretch-shortening cycle of the muscle-tendon complex, enhancing elastic capacity and neuromuscular responsiveness. Therefore, these exercises are often referred to as reactive neuromuscular training [46]. The program combines plyometric jumps and landings with balance-enhancing movements, all performed on the affected extremity.
  The program consists of three main phases: a warm-up, the main training session, and a cool-down. The warm-up includes 5 minutes of slow jogging and 5 minutes of high-knee running. The main session involves progressively intensified combined balance and plyometric exercises. The cool-down includes 5 minutes of low-intensity running followed by static stretching exercises targeting lumbar extensors, hamstrings, quadriceps
  Interventions: Other: Exercise
- The stroboscopic group (Experimental): The stroboscopic group will perform all exercises wearing stroboscopic glasses (SENAPTEC, Beaverton, Oregon). These glasses use liquid crystal lenses that alternate between transparent and (nearly) opaque states via electric current.a mid-range opacity setting will be used to avoid extreme visual deprivation [50,51].
  Plyometric training emphasizes the stretch-shortening cycle of the muscle-tendon complex, enhancing elastic capacity and neuromuscular responsiveness. Therefore, these exercises are often referred to as reactive neuromuscular training [46]. The program combines plyometric jumps and landings with balance-enhancing movements, all performed on the affected extremity.
  The program consists of three main phases: a warm-up, the main training session, and a cool-down. Exercise volume, repetitions, and rest intervals are systematically planned. Each set is followed by 15-30 seconds of rest. Intensity progresses from low to moderate throughout the program.
  Interventions: Other: Exercise stroboscopic
- Control group (Other): The control group will continue with their routine training program and will not participate in any intervention.
  Interventions: Other: training

INTERVENTIONS:
Other: Exercise stroboscopic — In this study, balance and plyometric exercises will be performed by one group using stroboscopic glasses.
  Arms: The stroboscopic group
Other: training — routine training program
  Arms: Control group
Other: Exercise — balance and plyometric exercises
  Arms: The non-stroboscopic group

SUMMARY:
The aim of this study is to investigate the effects of an 8-week combined balance and plyometric exercise program using stroboscopic glasses on muscle morphology, dynamic balance, and proprioception in athletes with a history of ankle sprains. The primary objective is to assess the effectiveness of innovative rehabilitation strategies and their integration into clinical practice. Ultimately, the study seeks to accelerate recovery, reduce recurrence risk, and support long-term functional outcomes. Additionally, the findings are expected to fill current gaps in the literature on muscle architecture and performance, contributing scientifically to rehabilitation protocols.

Hypotheses:

Hypothesis 1: Stroboscopic visual feedback exercise training affects ankle muscle architecture in athletes.

Hypothesis 2: Stroboscopic visual feedback exercise training affects dynamic balance in athletes.

Hypothesis 3: Stroboscopic visual feedback exercise training affects ankle proprioception in athletes.

Hypothesis 4: Stroboscopic visual feedback exercise training affects postural stability in athletes.

DETAILED DESCRIPTION:
Ankle sprain, particularly injuries to the lateral ligament complex of the ankle joint, is one of the most common lower extremity injuries among athletes [1]. The prevalence of sports-related ankle injuries ranges between 20% and 50%, and according to the American Academy of Orthopaedic Surgeons, approximately 25% of athletic injuries are related to the foot and ankle. High-performance sports such as basketball, football, and volleyball, which involve running, jumping, and sudden directional changes, place significant mechanical load on the ankle, thereby substantially increasing the risk of injury [2].Numerous potential risk factors for the incidence and recurrence of lateral ankle sprains (LAS) have been identified in the literature. These include a history of prior sprains, gender, height, body weight, anatomical foot posture, malalignments such as genu varum and pes cavovarus, joint laxity, range of motion, muscle strength, proprioception, reaction time, and postural sway [5]. muscle strength, reaction time, and postural sway [8].

High rates of re-injury and long-term sequelae following ankle sprains have been documented. Previous studies have shown that at least 73% of individuals who experience recurrent ankle sprains develop residual symptoms such as pain, a sense of giving way, a lack of confidence in the ankle, loss of proprioception, and neuromuscular control deficits.These factors increase the risk of re-injury and the likelihood of developing chronic ankle instability (CAI) [9]. Although the mechanisms behind recurrent sprains are not fully understood, studies indicate decreased muscle activation post-injury, prolonged response times to perturbations, and altered activation onset of the evertor, plantar flexor, and dorsiflexor muscles. The primary clinical goal following a lateral ankle sprain (LAS) is to prevent recurrence [23]. In this regard, conservative treatment is considered the primary approach for symptom management and recurrence prevention. Understanding etiological factors, mechanisms, and triggers underlying recurrent LAS is crucial for designing effective rehabilitation exercises [24]. The ROAST consensus by the International Ankle Consortium underscores the importance of addressing mechanical and sensorimotor deficits following LAS [25].

Reduced somatosensory input at the ankle joint and increased reliance on visual cues are considered key contributors to the sensation of giving way and repeated sprains [26]. Such somatosensory changes can negatively impact joint position and movement sense, becoming critical injury risk factors. Although definitive strategies to modify motor cortex excitability are yet to be developed, interventions targeting these neural components are vital for optimal recovery and the prevention of somatosensory dysfunction [27]. Traditional rehabilitation approaches for recurrent sprains typically include strength, proprioception, and dynamic balance exercises. Balance training has long been a cornerstone of rehabilitation for individuals with chronic ankle instability (CAI), as it is believed to effectively enhance mechanoreceptor activity through stimulation of the ankle capsule and ligaments. This process enhances sensory output and activates gamma motor neurons during training [28,29]. Multimodal comprehensive exercise protocols are regarded as effective treatment options for individuals with CAI [30,31].

Integrating targeted rehabilitation interventions aimed at restoring proprioception, muscle strength, and neuromuscular control is essential for breaking the cycle of sensory and motor dysfunction. Recent studies support that combining proprioceptive and strengthening exercises improves functional stability and reduces recurrence risk [32]. However, earlier studies suggest traditional CAI interventions inadequately address post-sprain somatosensory deficits and fail to modify the increased reliance on visual cues in CAI patients [33,34]. Therefore, treatment strategies targeting neurophysiological dysfunctions may offer a promising approach in CAI rehabilitation. These interventions, focusing on somatosensory deficits, could provide a novel perspective in managing CAI and significantly enhance rehabilitation outcomes [33].

The effects of visual input on somatosensory function have gained attention in recent years. Stroboscopic visual training, involving intermittently disrupted visual feedback using specially designed glasses, is based on this principle [35]. These stroboscopic glasses alternate between transparent and opaque states every 100 milliseconds, reducing visual input and prompting the central nervous system to rely more heavily on somatosensory and vestibular information [36]. Such visual feedback tools offer a novel approach to proprioceptive training, enhancing neuromuscular and postural control [37]. Literature indicates that using these glasses significantly improves postural control in individuals with functional ankle instability following rehabilitation [35]. Stroboscopic glasses incorporated into proprioceptive exercises may help the central nervous system recalibrate proprioceptive input weighting, thereby enhancing the use of somatosensory and vestibular afferents for neuromuscular control [38]. This supports improved postural control and safer responses to perturbations in CAI patients [36].

Lee et al. investigated the effects of stroboscopic visual training on reweighting visual input in individuals with recurrent ankle sprains. The group using stroboscopic glasses showed improved eversion and dorsiflexion angles as well as increased activation in the tibialis anterior and peroneus longus muscles [39]. However, no study to date has explored the effects of these glasses on ankle muscle architecture in individuals with recurrent sprains.

Currently, there is no comprehensive study examining the changes in muscle architecture and performance around the ankle in athletes with recurrent ankle sprains. This underscores the need for in-depth investigation into these changes and their impact on ankle stability. The aim of this study is to investigate the effects of an 8-week combined balance and plyometric exercise program using stroboscopic glasses on muscle morphology, dynamic balance, and proprioception in athletes with a history of ankle sprains. The primary objective is to assess the effectiveness of innovative rehabilitation strategies and their integration into clinical practice. Ultimately, the study seeks to accelerate recovery, reduce recurrence risk, and support long-term functional outcomes. Additionally, the findings are expected to fill current gaps in the literature on muscle architecture and performance, contributing scientifically to rehabilitation protocols.

ELIGIBILITY:
Inclusion Criteria:

1. At least 5 years of active participation in any sports branch.
2. At least two significant LAS incidents associated with inflammatory symptoms (pain, swelling).
3. Most recent sprain occurred at least 3 months before study commencement.
4. Feeling of ankle giving way at least twice in the past 6 months.
5. No history of surgical intervention affecting lower extremity sensorimotor function and no history of ankle fractures.
6. Cumberland Ankle Instability Tool (CAIT) score ≤25.
7. Foot and Ankle Ability Measure (FAAM) score below 90%.
8. FAAM Sports subscale score below 80%.

Exclusion Criteria:

1. History of any ankle fracture.
2. Surgical intervention or systemic disease affecting lower extremity sensorimotor function.
3. History of neurological disorders.
4. Acute musculoskeletal injury to the lower extremity within the last month.
5. Visual or vestibular disorders affecting balance or coordination.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Muscle Architecture Assessment | 1 hour
  Muscle architectural variables will be assessed using an HS60 (Samsung Medicine, Gangwon-do, Korea) ultrasound system equipped with a 5-13 MHz linear probe. Muscle cross-sectional area (MCA) measurements of the ankle circumference muscles will be performed under two different conditions, resting and maximal voluntary contraction (MVC), using the B-mode (brightness mode) ultrasound method. All measurements will be completed under these two conditions. Ultrasound imaging procedures will be performed by a researcher physical therapist experienced in musculoskeletal ultrasound.
Dynamic Balance Assessment | 15 minute
  The Y balance test, a short and practical variation of the star balance test, will be used to assess dynamic stability. Athletes will perform the Y balance test according to the test procedures defined by Plisky et al. Three white bands, each 125 cm in length, will be affixed to the ground to form a Y shape, with the small angle at 90° and the two larger angles at 135°, and centimeter-scale markings will be added to the bands by hand.Participants will be positioned at the center of the apparatus with the second phalanges of the extremity being tested in the coronal plane and the metatarsophalangeal joints in the sagittal plane, both aligned with the midline. Participants will be asked to stand with their hands at the level of the iliac crest, adjacent to their bodies, and with the foot to be measured on the ground, to reach out with the other foot in the anterior, posteromedial, and posterolateral directions, once in each direction, and to lightly touch the final point they can reach.
Proprioception Assessment | 15 minute
  An ankle joint position sense test will be administered to assess deficiencies in ankle proprioception. An electronic goniometer will be used to assess ankle joint position sense. The reliability of this test among recreational athletes with ankle instability has been reported as ICC = 0.94-0.98 [45].
  Athletes will be seated with their knees flexed at 90°, and their eyes will be closed to eliminate visual cues. The ankle subtalar joint (STJN) will be held in a neutral position, and the goniometer will be set to zero. The ankle will be passively moved through 10° dorsiflexion, 10° eversion, 15° plantar flexion, or 15° inversion, and then returned to the neutral position [46]. Participants will then be asked to actively perform these movements as closely as possible to the previous movements. Three repeated measurements will be taken for each test angle, and deviations from the target angle will be recorded.
Postural Stability Assessment | 20 minute
  Athletes' postural stability and center of pressure (CoP) assessments will be performed using the Prokin force platform (Prokin PK 252). The Prokin PK 252 is a proprioceptive system used for static and dynamic balance assessment and training. In this study, the "Static and Dynamic Stability Assessment Program" will be used to provide detailed and accurate data on participants' static standing posture through the stabilometry platform and sensors placed on the body [47]. During the test, participants' standing position will be determined with their feet shoulder-width apart, and their foot positions will be aligned at equal distances from the origin point, using the lines on the platform's x and y axes as references.First, a single-leg static stability test will be performed. This test will be administered in two sub-tests: with eyes open and with eyes closed.

SECONDARY OUTCOMES:
Foot and Ankle Ability Measure (FAAM) | 15 minute
  Athletes' physical functions will be assessed using the Turkish version of the Foot and Ankle Ability Measure (FAAM). FAAM is a self-report measurement tool developed to assess the physical functions of individuals with musculoskeletal problems related to the foot and ankle. The FAAM consists of a total of 29 items, including a 21-item Activities of Daily Living (ADL) subscale and an 8-item Sports subscale. The Sports subscale provides a sports-specific subclass to assess the ability to perform sports-related activities. Each question is scored using a 5-point Likert scale ranging from 0 (unable to perform) to 4 (able to perform without difficulty). The maximum score for the ADL subscale is 84, while the maximum score for the Sports subscale is 32. Total scores are calculated as percentage scores ranging from 0% to 100%, with a higher score indicating a higher level of function [48].
Cumberland Ankle Instability Tool (CAIT) | 10 minute
  Cumberland Ankle Instability Tool Developed in 2006, the Cumberland Ankle Instability Tool 17 (CAIT) was the first to provide a numerical value measuring the level of ankle instability based on individuals' perceptions [41].
  The CAIT scale, designed to assess functional ankle instability levels, consists of 9 questions; the maximum total score is 30 and the minimum is 0. A lower total score indicates more severe functional ankle instability. Test-retest reliability was found to be excellent at 0.96. The CAIT is the first tool to validly and reliably assess functional ankle instability. In the study, the cutoff score was set at 27.5, with a sensitivity of 82.9% and a specificity of 74.7%. Finally, the CAIT score has the potential to predict the risk of re-sprain in individuals with functional ankle instability. Individuals with a sprained ankle and a low CAIT score have a higher likelihood of re-sprain, while those with a high CAIT score have a lower likelihood of re-sprain [42].

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided